CLINICAL TRIAL: NCT00254306
Title: Functional Brain Imaging in Recreational Users of Ecstasy
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Aviv Weinstein, Hadassah Medical Organization
Other Study IDs: 050893-HMO-CTIL; n/q
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Amphetamine-Related Disorders
Keywords: Ecstasy; D2 Dopamine Receptor; IBZM; MDMA
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: ex-"ecstasy" users
- 2: control subjects

SUMMARY:
Recreational use of "ecstasy" (MDMA; 3,4-methylenedioxymethamphetamine) is associated with long-lasting effects on metabolism in the human brain. The investigators propose to investigate whether chronic use of "ecstasy" is associated with impairment in motor skills and function of the dopaminergic system in recreational users of "ecstasy" compared with healthy volunteers. This will be done by scanning control subjects and "ecstasy" users at baseline and after performing on a motorbike riding computer game, while imaging dopamine in vivo with I123-IBZM (a D2 receptor radiotracer), using single photon emission computed tomography (SPECT).

DETAILED DESCRIPTION:
Recreational use of "ecstasy" (MDMA; 3, 4-Methylenedioxymethamphetamine) is associated with long-lasting effects on metabolism in the human brain. In particular, there is evidence of long-term damage to the brains' neurotransmitter serotonin (5-HT). It is also known that chronic use of Methamphetamine (which is similar in its chemical structure to "ecstasy") is linked to impaired cognitive and motor skills despite recovery of dopamine transporters (DAT). We have investigated whether chronic use of "ecstasy" is causing any impairment in motor skills and function of the dopaminergic system in recreational users of "ecstasy". In our preliminary study, we have scanned control subjects and "ecstasy" users, at baseline and after performing on a motorbike riding computer game while imaging dopamine in vivo with [123I] IBZM (a D2 receptor radiotracer) in Single Photon Emission Computed Tomography (SPECT). We showed:

1. Lower measures of D2 at baseline in ecstasy users compared with control subjects, that means lower level of dopaminergic activity in "ecstasy" users.
2. Significant displacement of [123I] IBZM by endogenous dopamine released during the game in healthy subjects unlike "ecstasy" users, that means that recreational users of "ecstasy" release much less natural dopamine.
3. No difference between the groups in performance (reaction time) on riding the game after a year of recovery.

Our results show preliminary evidence for dopaminergic deficiency in "ecstasy" users, a finding that has not been shown before. However, similar to other drugs of abuse, it is not known whether dopaminergic deficiency is the cause or consequence of the use of "ecstasy". We now propose to proceed to scan more recreational users of "ecstasy" in order to assess whether chronic use of "ecstasy" is associated with deficient dopaminergic neurotransmission in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic users of ecstasy, and healthy controls, with no other diseases or drug abuse

Exclusion Criteria:

* Pregnant and breast feeding women
* Aged below 18
* Neurological disorders
* Drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from treatment centers for drug abuse. Control subjects will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yodphat Krausz, MD, Principal Investigator — Hadassah Medical Organization; Aviv M Weinstein, Ph.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Dept. of Nuclear Medicine, Hadassah Hospital, Ein Kerem, Jerusalem, Israel